CLINICAL TRIAL: NCT07185295
Title: Short-term Interruption Versus Continuous Anticoagulation in Colorectal Polypectomy, a Randomized Multicenter Investigator-initiated Non-inferiority Clinical Trial
Brief Title: Short-term Interruption Versus Continuous Anticoagulation in Colorectal Polypectomy
Acronym: POLYPHEM
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Outcomes'10 (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECA-HRC-POLYPHEM-04
Record Dates: First submitted 2025-09-05; First posted 2025-09-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Anticoagulated Patients
Keywords: Anticoagulant therapy; colorectal polypectomy; Oral anticoagulants; colonoscopy; Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: The intervention consists of managing anticoagulation in two different ways during colorectal polypectomy: Comparison of Temporary Interruption of Anticoagulation (Standard of Care) vs. Continuation of Anticoagulation (Interventional Arm)
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maintained Anticoagulant Therapy (Experimental): Patients in this treatment group will continue their anticoagulant therapy during the procedure. For those on vitamin K antagonists (VKAs), INR levels will be checked 7-14 days before the endoscopy, and doses adjusted if necessary to maintain therapeutic range (<3.5) before the procedure. Patients on direct oral anticoagulants (DOACs) will skip only the morning dose on the day of the procedure without other changes.
  Interventions: Procedure: To maintain anticoagulant therapy during the polypectomy of colorectal lesions
- Discontinued Anticoagulant Therapy (No Intervention): In patients assigned to this treatment arm, anticoagulation will be temporarily discontinued following the recommendations of the 2021 BSG-ESGE clinical practice guideline. The distinction between high and low thrombotic risk will be made according to guidelines.

INTERVENTIONS:
Procedure: To maintain anticoagulant therapy during the polypectomy of colorectal lesions — Group A
  Arms: Maintained Anticoagulant Therapy

SUMMARY:
This study is designed to find out if it is safe to keep taking blood-thinning medicine during the removal of polyps from the colon or rectum.

It includes patients who regularly take blood thinners and need an elective colonoscopy.

The main goal is to see how often patients have serious bleeding after the polyp removal within 30 days.

The study is being done in several hospitals, and doctors evaluating the results do not know which treatment patients receive.

DETAILED DESCRIPTION:
This multicenter, phase IV, assessor-blinded, non-inferiority clinical trial evaluates the safety of maintaining oral anticoagulant therapy during colorectal polypectomy. The study population includes patients receiving chronic oral anticoagulation treatment with vitamin K antagonists (VKAs) or direct oral anticoagulants (DOACs) who are scheduled for elective colonoscopy for any indication.

The primary objective is to assess the incidence of clinically significant post-polypectomy bleeding within 30 days after the procedure. The trial tests the hypothesis that continuing anticoagulant therapy during polypectomy is non-inferior to interrupting it, with a non-inferiority margin set at 10%.

A total of 481 patients will be enrolled, with 241 patients per group. The intervention consists of maintaining ongoing anticoagulant treatment without modification before the procedure. This trial is classified as a low-intervention study according to regulatory guidelines and aims to provide evidence to optimize the management of anticoagulated patients undergoing colorectal polypectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Patients scheduled for elective outpatient colonoscopy for any indication, in whom removal of colorectal polyps will be performed if identified during the procedure.
* Anticoagulant treatment with vitamin K antagonists (acenocoumarol or warfarin) or direct oral anticoagulants (dabigatran, edoxaban, apixaban, or rivaroxaban) prior to the colonoscopy.

Exclusion Criteria:

* Concomitant antiplatelet therapy.

Age over 85 years.

Urgent colonoscopy.

Labile INR (time in therapeutic range less than 60%) documented in the previous 3 months in patients receiving VKAs.

Supratherapeutic INR (>3.5) at the time of the procedure in patients on VKAs.

Pregnancy.

Decompensated liver cirrhosis.

Inability, at the investigator's discretion, to understand the periprocedural anticoagulation regimen.

Known coagulopathy or bleeding diathesis, including platelet count <50,000/µl in the previous 12 months.

Scheduled endoscopic dilation.

Severe psychiatric disorder.

Removal of colorectal lesions by endoscopic submucosal dissection.

Previous diagnosis of renal failure defined as creatinine >2 mg/dl or clearance <30 ml/min.

Planned high bleeding risk procedure during simultaneous gastroscopy.

Previous inclusion in the trial. Patients may only be included once.

Patients who are not candidates for a second endoscopic intervention due to clinical conditions.

Any clinical situation or concomitant treatment that, in the investigator's opinion, poses a significant bleeding risk.

Patients with polyps larger than 4 cm pending endoscopic resection.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinically significant intraprocedural bleeding | 1 month
  Major bleeding during colonoscopy that requires procedure interruption, a drop in hemoglobin >2 g/dL, blood transfusion, interventional radiology, hospitalization, surgery, or results in death.
  The following data will be collected for bleeding events:
  * Date of the event.
  * Length of hospital stay: Quantitative nominal variable. Unit: days.
  * ICU admission: Binary variable (Yes/No).
  * Severity: Assessed according to the ASGE classification.
Clinically significant delayed hemorrhage | 1 month
  Gastrointestinal bleeding occurring within 30 days after completion of the colonoscopy that requires an emergency visit, hospitalization, or an intervention.
  Date of the event. - Length of hospital stay: Quantitative nominal variable. Unit: days. - ICU admission: Binary variable (Yes/No). - Severity: Assessed according to the ASGE classification.

SECONDARY OUTCOMES:
Acute Myocardial Infarction | 1 month
  A clinical syndrome characterized by evidence of myocardial necrosis in a clinical setting consistent with acute myocardial ischemia.
  Data collected will include event date, hospital stay duration, and ICU stay duration.
Hospitalization for Unstable Angina | 1 month
  Unscheduled hospitalization for the treatment of unstable angina occurring within 24 hours from symptom onset. Hospitalization is defined as admission to an inpatient unit or an emergency department visit resulting in a stay of at least 24 hours. Data collected will include event date, hospital stay duration, and ICU stay duration.
Deep Vein Thrombosis | 1 month
  Any deep vein thrombosis diagnosed in the upper body (internal jugular, subclavian, axillary/brachial) or lower extremities (iliac, femoral/popliteal, gastrocnemius, peroneal, posterior tibial), or in the inferior vena cava or deep splanchnic veins, as confirmed by ultrasound or contrast imaging techniques including computed tomography (CT), angiography, or magnetic resonance imaging (MRI). Data collected will include event date, hospital stay duration, and ICU stay duration.
Pulmonary Embolism | 1 month
  Any pulmonary embolism diagnosed by computed tomography (CT), ventilation-perfusion (V/Q) scan, invasive pulmonary angiography, echocardiography (thrombus visualized in the main pulmonary artery), or confirmed by autopsy. Data collected will include event date, hospital stay duration, and ICU stay duration.
Stroke, Including Transient Ischemic Attack | 1 month
  Stroke is defined as an acute episode of focal or global neurological dysfunction caused by a cerebral, spinal, or retinal vascular injury as a result of hemorrhage or infarction.
  Transient ischemic attack (TIA) is defined as a temporary (< 24 hours) episode of focal neurological dysfunction caused by cerebral, spinal, or retinal ischemia without acute infarction. Data collected will include event date, hospital stay duration, and ICU stay duration.
Peripheral Arterial Embolism or Thrombosis | 1 month
  Any embolism or arterial thrombosis diagnosed by computed tomography (CT), ultrasound, or magnetic resonance imaging (MRI) involving the splanchnic circulation, upper or lower extremities, or renal arteries. Data collected will include event date, type, hospital stay duration, and ICU stay duration.
Clinically non-significant intraprocedural bleeding | 1 month
  Bleeding that persists for more than 1 minute, requires endoscopic treatment, and does not meet the criteria for clinically significant intraprocedural bleeding.
Death | 1 month
  It will be recorded as a nominal categorical variable:
  - No/death If death is selected: Cause/unknown cause. It will be also recorded the date of death

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Clínica Rotger Quirónsalud, Palma, Balearic Islands
  - Servicio de Aparato Digestivo. Hospital Sierrallana. Barrio Ganzo,, Torrelavega, Cantabria
  - Servicio de Gastroenterología y Hepatología. Hospital Universitario Río Hortega., Valladolid, Castille and León
  - Servicio de Digestología, Hospital del Mar. Instituto Hospital del Mar de Investigaciones Médicas., Barcelona, Catalonia
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - Servicio de Gastroenterología. Hospital Universitario Príncipe de Asturias. Madrid., Alcalá de Henares, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Servicio de Gastroenterología y Hepatología. Unidad de Endoscopias. Hospital Universitario Puerta De Hierro., Majadahonda, Madrid
  - Servicio de Gastroenterología y Hepatología. Hospital Universitario San Agustín., Avilés, Principality of Asturias
  - Servicio de Aparato Digestivo. Hospital Universitario de Cabueñes, Oviedo, Principality of Asturias

IPD SHARING:
Plan to Share IPD: No